CLINICAL TRIAL: NCT05773027
Title: Integrated Alcohol and Sexual Assault Intervention for College Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lifespan (Other)
Responsible Party: Principal Investigator, Lindsay Orchowski Ph.D., Associate Professor (Research), Lifespan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R34AA020852 (NIH)
Record Dates: First submitted 2023-02-22; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Alcohol Drinking; Sexual Assault
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sexual Assault and Alcohol Feedback and Education (SAFE) (Experimental): SAFE includes a motivational interviewing session addressing alcohol use and risk for sexual aggression, a workshop addressing alcohol use and sexual aggression, and a booster session review.
  Interventions: Behavioral: SAFE
- Mindfulness-Based Control Condition (Active Comparator): The program includes the same amount of contacts as SAFE, including an individual session focused on mindfulness and stress, a group session, and a booster session review.
  Interventions: Behavioral: Mindfulness-Based Control Condition

INTERVENTIONS:
Behavioral: SAFE — SAFE includes a motivational interviewing session addressing alcohol use and risk for sexual aggression, a workshop addressing alcohol use and sexual aggression, and a booster session review.
  Arms: Sexual Assault and Alcohol Feedback and Education (SAFE)
Behavioral: Mindfulness-Based Control Condition — The program includes the same amount of contacts as SAFE, including an individual session focused on mindfulness and stress, a group session, and a booster session review.
  Arms: Mindfulness-Based Control Condition

SUMMARY:
This research will evaluate a new intervention that integrates evidence-based alcohol intervention strategies and promising sexual assault prevention strategies with the goal of decreasing sexual aggression among men who report heavy drinking; a particularly high risk group. Specifically, this study will conduct a randomized controlled pilot trial with college men who report heavy drinking to demonstrate the feasibility and acceptability of the proposed intervention. The main questions the study will answer are: 1) what is the feasibility of the recruitment plans, research design, intervention training methods, and delivery of the program?; and 2) does the intervention, relative to a mindfulness-based control condition, produce reductions in the quantity and frequency of alcohol use, perpetration of sexual aggression, and attitudes associated with sexual aggression over the 2- and 6-month follow-up. Follow-up assessments are completed at 2- and 6-months following the program. The intervention is compared to the mindfulness-based control group.

ELIGIBILITY:
Inclusion Criteria:

* Engaging in binge drinking, defined as 5 or more drinks per day for men on the same occasion by the Substance Abuse and Mental Health Services Administration on two or more occasions in the past month.
* Engaging in oral, vaginal, or anal sexual intercourse with a female partner one or more times in the past four months

Exclusion Criteria:

* Displaying symptoms consistent with alcohol use withdrawal
* Reporting current suicidal or homicidal ideation
* Meeting criteria consistent with a diagnosis of Antisocial Personality Disorder

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-identify as male.
Enrollment: 115 (Actual)
Dates: Start 2013-10-17 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
Alcohol use, heavy drinking quantity | Change from baseline alcohol use at 6 months.
  Number of heavy drinking days in the past month (Minimum = 0, Maximum = 31), assessed via the timeline follow-back. Greater scores mean worse outcomes.
Alcohol use, drinks per week | Change from baseline alcohol use at 6 months.
  The average number of drinks per week (Minimum = 0, Maximum = unspecified), assessed via the timeline follow-back. Greater scores mean worse outcomes.
Sexual aggression perpetration | Change in severity and frequency in comparison to control at 6-months.
  Assessed via the sexual experiences survey. Scored based on frequency and severity (Minimum = 0, Maximum = 63). Higher scores mean worse outcomes.

SECONDARY OUTCOMES:
Protective behavioral strategies | Change in protective behavioral strategy use in comparison to control at 6-months.
  Assessed via the Self Control Questionnaire (Minimum = 37, Maximum = 185). Higher scores mean more positive outcomes.
Perceived peer drinking norms | Change in perceived peer norms relative to control at 6-months.
  Assessed via the drinking norms rating form (Minimum = 0, Maximum = unspecified). Higher scores mean worse outcomes.
Perceived peer norms regarding sexual aggression: Perceived peer bystander intervention | Change in perceived peer bystander intervention in comparison to control at 6-months.
  Assessed via the sexual social norms inventory, perceived peer bystander intervention (Minimum = 8, Maximum = 40, higher scores better outcomes).
Perceived peer norms regarding sexual aggression: Perceived peer engagement in sexual coercion | Change in perceived peer engagement in comparison to control at 6-months.
  Assessed via the sexual social norms inventory, regarding perceived peer engagement in sexual coercion (Minimum = 7, Maximum = 35, lower are better outcomes).
Perceived peer norms regarding sexual aggression: Peer comfort with sexual aggression | Change in peer comfort with sexual aggression relative to control at 6-months.
  Assessed via the sexual social norms inventory, perception of peer comfort with sexual aggression (Minimum = 7 , Maximum = 35, lower are better outcomes).
Attitudes relating to sexual aggression: Rape myth acceptance | Change in rape myth acceptance relative to control at 6-months.
  Assessed via the rape myth acceptance scale (Minimum = 7, Maximum = 140, higher are worse outcomes).
Attitudes relating to sexual aggression: Hyper gender ideology | Change in hyper gender ideology and increases relative to control at 6-months.
  Assessed via the hyper gender ideology scale (Minimum = 19, Maximum = 114, higher scores are worse outcomes).
Attitudes relating to sexual aggression: Labeling of consent | Change in labeling of consent relative to control at 6-months.
  Assessed via the labeling of consent scenarios (Minimum = 1, Maximum= 10, higher scores are better outcomes).
Bystander intervention intention to help strangers | Change in intention to help strangers relative to control at 6-months.
  Assessed via the intentions to help strangers scale (Minimum = 0, Maximum = 800, higher scores are better outcomes).
Bystander intervention intention to help friends | Change in intent to help friends relative to control at 6-months.
  Assessed via the bystander intentions to help friends scale (Minimum = 0, Maximum = 1000, higher scores are better outcomes).
Bystander intervention attitudes | Change in bystander attitudes relative to control at 6-months.
  Assessed via the bystander attitudes scale (Minimum = 51, Maximum = 255, higher scores are better outcomes).

OTHER OUTCOMES:
Motivation to change | Change in motivation relative to control from baseline to immediately after the session.
  Assessed via the Contemplation latter (Minimum = 0, Maximum = 10, higher scores are better outcomes).
Self-Efficacy | Change in self-efficacy relative to control at from baseline to immediately after the session.
  Assessed via the brief situational confidence questionnaire (Minimum = 0, Maximum = 100, higher scores are better outcomes).
Drinking intentions | Change in drinking intentions relative to control from baseline to immediately after the session.
  Assessed via the drinking intention weekly report (Minimum = 0, Maximum = Unspecified, higher scores are worse outcomes).

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing requests can be made by contacting the study PI.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data can be requested from the PI .
Access Criteria: A data sharing agreement can be requested by contacting the PI.

REFERENCES:
- [Derived] Orchowski LM, Merrill JE, Oesterle DW, Barnett NP, Borsari B, Zlotnick C, Haikalis MP, Bekowitz AD. Integrated Alcohol Use and Sexual Assault Prevention Program for College Men Who Engage in Heavy Drinking: Randomized Pilot Study. JMIR Form Res. 2023 Nov 23;7:e47354. doi: 10.2196/47354. PMID 37995129